CLINICAL TRIAL: NCT01900379
Title: Impact of the Obstructive Sleep Apnea Syndrome Treatment and Ventricular Function in Heart Failure Patients Undergoing Coronary Artery Bypass Surgery or Other Coronary Reperfusion
Brief Title: PAC-IC-SAOS Obstructive Sleep Apnea Syndrome and Ventricular Function
Acronym: PAC-IC-SAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1310; 2013-A00543-42 (Other: ANSM)
Record Dates: First submitted 2013-07-05; First posted 2013-07-16 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure; Arteriosclerosis of Coronary Artery Bypass Graft or Other Coronary Reperfusion; Sleep Apnea, Obstructive
Keywords: Obstructive sleep apneas syndrome; Continuous positive airway pressure treatment; Heart failure; Coronary reperfusion surgery
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OSA/CPAP (Experimental): OSA patients intervention : CPAP treatment
  Interventions: Procedure: CPAP treatment
- OSA/sham CPAP (Sham Comparator): OSA patients intervention : Sham CPAP treatment
  Interventions: Other: Sham CPAP treatment
- control group (No Intervention): Patients without any apnea syndrome

INTERVENTIONS:
Procedure: CPAP treatment — This device consists in a nasal continuous positive airway pressure. It will be applied just after CABG and for 3 months for OSA/CPAP patients group.
  Arms: OSA/CPAP
Other: Sham CPAP treatment — This device consists in a sham continuous positive airway pressure. It will be applied just after CABG and for 3 months for OSA/sham CPAP patients group.
  Arms: OSA/sham CPAP

SUMMARY:
The aim of this clinical trial is to evaluate the effect of obstructive sleep apnea syndrome (OSAS) treatment in heart failure patients following coronary artery bypass graft (CABG) surgery or other coronary reperfusion.

DETAILED DESCRIPTION:
This clinical trial is a double-blind, randomized, placebo-controlled study.

The first objective is to evaluate the influence of continuous positive airway pressure (CPAP) treatment for OSAS on the ventricular function improvement in heart failure patients, in comparison with OSA patients treated with sham CPAP. This treatment will be instaurated just after the coronary reperfusion surgery

Secondary objectives :

* Evaluation of the effect of CPAP treatment on the endothelial function
* Evaluation of the effect of CPAP treatment on systemic inflammation
* Evaluation of the effect of CPAP treatment on oxidative stress,
* Evaluation of the effect of CPAP treatment on insulin resistance,

after the coronary reperfusion surgery, in comparison with OSA patients treated with sham CPAP and non apneic control patients, with heart failure.

* Assessment of the impact of nocturnal desaturation level on the vascular reactivity and atherosclerosis of mammary vessels collected during surgery.
* Assessment of the impact of nocturnal desaturation level on the oxidative stress, inflammation and insulin sensitivity on abdominal and epicardiac adipose tissue collected during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Bypass Surgery or other coronary reperfusion
* Heart failure patient: with altered left ventricular ejection fraction by ultrasonography (≤ 50% in 2D) or in 3D

Exclusion Criteria:

* Aortic or mitral valvular replacement
* Aortic surgery
* Triple stimulator implanted less than 6 months ago
* Patient already treated for a SAOS syndrome
* Patient with a central sleep apnea syndrome
* Patient with malignant evolutive pathology
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Percent of ventricular function recovery (left ventricular ejection fraction (LVEF)) improvement conferred by CPAP post-operative treatment | After 3 months of CPAP post-operative treatment
  Measurement of the left ventricular ejection fraction by a cardiac ultrasonography

SECONDARY OUTCOMES:
Assessment of CPAP effect on the endothelial function, after the surgery in comparison with sham CPAP treated patient with heart failure and OSAS. | After 3 months of CPAP post-operative treatment
  Measurement of peripheral arterial tone
Assessment of CPAP effect on the endothelial function, after the surgery in comparison with sham CPAP treated patient with heart failure and OSAS. | After 3 months of CPAP post-operative treatment
  Measurement of pulse wave velocity
Assessment of the impact of nocturnal desaturation level on the vascular atherosclerosis of mammary vessels collected only during CABG surgery. | Sleep disordered breathing level, 2 months before surgery
  By immunological and histological analysis of mammary vessels
Assessment of the impact of nocturnal desaturation level on the oxidative stress, inflammation and insulin sensitivity of the abdominal and epicardiac adipose tissue collected during surgery. | Sleep disordered breathing level, 2 months before surgery
  Measuring inflammatory and oxidative adipose markers
Assessment of the impact of nocturnal desaturation level on the vascular reactivity of mammary vessels collected during surgery. | Sleep disordered breathing level, 2 months before surgery
  By immunological and histological analysis of abdominal and epicardiac adipose tissue
Assessment of CPAP effect on the systemic inflammation and oxidative stress, the insulin resistance, after the surgery in comparison with sham CPAP treated patients with heart failure and OSAS. | After 3 months of CPAP post-operative treatment
  Measurement of inflammatory and oxidative serum markers

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, MD, PhD, Principal Investigator — University Hospital of Grenoble, France
Locations (1):
- University Hospital of Grenoble, Grenoble, France